CLINICAL TRIAL: NCT00783991
Title: Investigating the Impact of Mode of Administration on Item Response
Status: Completed | Type: Observational
Sponsor: Stony Brook University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); QualityMetrics (Industry); Endeavor Health (Other); Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 07-05; 5U01AR052170-02 (NIH)
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Depression; Rheumatoid Arthritis
Keywords: IVF; PDA; PC; CAT; COPD; MDD; RA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Depression; Arthritis, Rheumatoid

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- IVR-PC: This group will have instruments administered through interactive voice response (IVR) and personal computer (PC).
- PP-PC: This group will have instruments administered through paper and pencil (PP) and PC.
- PDA-PC: This group will have instruments administered by personal digital assistant (PDA) and PC.
- PC-PC: This group will have all instruments administered through PC.

SUMMARY:
The Patient-Reported Outcomes Measurement Information System (PROMIS) is an NIH Roadmap initiative to develop a computerized system measuring patient-reported outcomes in respondents with a wide range of chronic diseases and demographic characteristics. In the first four years of its existence, the PROMIS network developed item banks for measuring patient-reported outcomes in the areas of pain, fatigue, emotional distress, physical function, and social functioning. During the item banking process, the PROMIS network conducted focus groups, individual cognitive interviews, and lexile (reading level) analyses to refine the meaning, clarity, and literacy demands of all items. The item banks were administered to over 20,000 respondents and calibrated using models based on item response theory (IRT). Using these IRT calibrations, computerized adaptive test (CAT) algorithms were developed and implemented. The network has designed a series of studies using clinical populations to evaluate the item attributes, examine their utility as CATs, and validate the item banks. More information on the PROMIS network can be found at www.nihpromis.org.

This study is designed to examine how differences in modes of data capture affect psychometric properties and score differences and to evaluate the consistency of these results across three PROMIS health domains: emotional distress-depression, fatigue, and physical function. Four modes of administration will be compared: interactive voice response (IVR) technology, paper and pencil questionnaire, personal computer, and personal digital assistant (PDA). A total of 800 patients will be enrolled from three diagnostic groups: chronic obstructive pulmonary disease (COPD), depression, and rheumatoid arthritis. The study will test for equivalence across modes of administration, with the hypothesis that there are no mode effects; if mode effects are found, their magnitude across modes will be estimated. This network project will result in an improved understanding of the effect of assessment mode on patient-reported outcome (PRO) data. Guidance from this project can help in planning future PROMIS activities beyond the present PROMIS program.

DETAILED DESCRIPTION:
This study is designed to systematically test the impact of mode of administration on patient-reported outcomes measures included in the PROMIS item banks. It is designed as a randomized cross-over study. Two non-overlapping alternate forms (Form A [FA] and Form B [FB]) with eight unique items each from three of the PROMIS domains (emotional distress-depression, fatigue, physical function) will be developed. Respondents will answer one of the forms by automated phone interview using interactive voice response (IVR) technology, paper and pencil questionnaire (PP), personal computer (PC), or personal digital assistant (PDA) technology. The other form will always be answered by PC. The order in which the forms are administered will be randomized. The two assessments will be separated by a short interval (e.g., 5 to 10 minutes), but will take place on the same day. The study is powered to evaluate equivalence within a score difference of +/-2.0 on a T-score metric (standard deviation of 10) with 85% power. Data for the IVR-PC, PP-PC, and PC-PC modes will be collected via Polimetrix (n=200 per arm, with random assignment to arm); data for the PDA-PC mode will be collected via Stony Brook (n=200). Respondents will have one or more of the chronic conditions studied in other Wave 2 studies (COPD, depression, or rheumatoid arthritis).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis given by treating physician
* Respondents required to take one or more of the following medications for their treatment:

  1. COPD: Inhalative steroids (e.g., budesonide, beclometasone), oral medication with theophylline (dimethylxanthine), 2 mimetic (e.g., formoterol, salmeterol), leukotriene antagonists (e.g., montelukast), or oral corticosteroids (e.g., prednisolone)
  2. DEP: Anti-depressive drugs (e.g., mirtazapine, escitalopram) and/or received a recognized psychotherapeutic treatment for depression within the last year
  3. RA: Anti-inflammatory medications (e.g., Cox-2 inhibitors, acetylsalicylic acid of more than 500mg/d, diclofenac, ibuprofen), immunosuppressants (e.g., methotrexate, leflunomide), immune modulators (e.g., infliximab, etanercept), or steroids (e.g., prednisolone) for current treatment of RA
* Fluent in English
* Have Internet access and an e-mail address (for the IVR-PC, PP-PC and PC-PC arms)
* Willing and able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community samples with at least one of these conditions: chronic obstructive pulmonary disease (COPD), depression (DEP), or rheumatoid arthritis (RA).
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
IRT-derived scores from two parallel static short forms containing eight items each from three PROMIS domains (emotional distress-depression, fatigue, physical function) | One time assessment
Respondent preference and satisfaction with mode of administration | One time assessment

CONTACTS AND LOCATIONS:
Overall Officials: John E. Ware, PhD, Principal Investigator — QualityMetrics; Arthur Stone, PhD, Principal Investigator — Stony Brook University
Locations (2):
- United States (2):
  - Polimetrix, Palo Alto, California
  - Rheumatology Associates of Long Island, Smithtown, New York